CLINICAL TRIAL: NCT02235896
Title: Cardiovascular Disease Prevention Among African-Americans by FAITH! (Fostering African-American Improvement in Total Health)
Brief Title: Reducing CVD Risk in African Americans Faith Communities
Acronym: FAITH!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sharonne Hayes, Professor of Medicine, Cardiovascular Diseases, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14-004122
Record Dates: First submitted 2014-09-05; First posted 2014-09-10 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Cardiovascular Disease Risk Factors
Keywords: risk factors, African American, lipids, blood pressure
MeSH Terms: interventions — Educational Status; Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Education/Behavior Modification (Other): Education/Behavior modification program
  Interventions: Behavioral: Education/Behavior Modification

INTERVENTIONS:
Behavioral: Education/Behavior Modification — Education, lifestyle counseling, experiential cooking, exercise classes.

SUMMARY:
The ultimate goal of our partnership with local African-American churches is to implement an effective, multi-component intervention to increase awareness of the critical importance of healthy lifestyle in the prevention of cardiovascular disease (CVD). We will utilize the American Heart Association (AHA) prevention strategy, "Life's Simple 7" to address the major risk factors for CVD: diet, smoking, physical inactivity, hypertension, diabetes, cholesterol and obesity in order to improve overall cardiovascular health. Our main strategy consists of a community-based participatory research approach that involves focus groups to assess participant knowledge and beliefs about CVD risk factors prior to program initiation. We will also determine participant dietary and exercise practices, knowledge and perceptions related to healthy lifestyle and chronic diseases, demographic/health status information, health care utilization, biometrics (weight, blood pressure, blood tests for glucose and cholesterol, etc.) and attitudes about medical research at baseline, program completion and 6-month follow-up.

DETAILED DESCRIPTION:
Church goers will undergo, baseline assessment of knowledge attitudes and behavior survey as it relates to CVD risk and anthropomorphic measurements. A 3 month experiential educational program will be provided at 2 locations. At 6 months after baseline a followup measure will be obtained

ELIGIBILITY:
Inclusion:

* Age >18 yrs,
* able to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Knowledge, attitudes about CVD and CVD risk | 1 year
  Change from baseline in knowledge and attitudes about CVD and CVD risk as measured by survey
Behavior change | 1 year
  Self reported diet composition, physical activity, smoking and stress

SECONDARY OUTCOMES:
CVD Risk factors | 1 year
  weight, lipids, blood glucose, BMI, Blood Pressure, % body fat, waist circumference
Attitudes about participation in Research | 1 year
  Knowledge and attitudes about medical research participation assessed by survey

CONTACTS AND LOCATIONS:
Overall Officials: Sharonne Hayes, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Brewer LC, Morrison EJ, Balls-Berry JE, Dean P, Lackore K, Jenkins S, Cohen C, Johnson J, Ellis F, Mangum DC, Hayes SN, Patten C. Preventing cardiovascular disease: Participant perspectives of the FAITH! Program. J Health Psychol. 2019 Oct;24(12):1710-1723. doi: 10.1177/1359105317695878. Epub 2017 Feb 1. PMID 28810418